CLINICAL TRIAL: NCT01106417
Title: Phase 2 Study Evaluating Safety and Preliminary Efficacy of NeoFuse When Combined With MasterGraft Matrix in Subjects Undergoing Multi-Level Anterior Cervical Discectomy and Fusion With Anterior Cervical Plate Fixation
Brief Title: Safety and Efficacy Study of NeoFuse in Subjects Undergoing Multi-Level Anterior Cervical Discectomy and Fusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSB-CF001
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Cervical Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: Cervical Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis; Stem cells; Adult Stem Cells; Anterior cervical discectomy and Fusion (ACDF); Anterior Cervical Plate Fixation
MeSH Terms: conditions — Spinal Stenosis | interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: Subjects received treatment in one of two parallel arms.
  Treatment Arm 1; NeoFuse (a biologic, consisting of STRO-3 immunological selected allogeneic Mesenchymal Precursor Cells, derived from adult bone marrow mononucleated cells) with Mastergraft Matrix (a medical device that is compression resistant and embedded with Mastergraft Granules). Subjects received 10 million Neufuse cells per treated cervical interbody level involved in the fusion. Either 2 or 3 levels were involved for a total of either 20 million or 30 million Neofuse cells.
  Treatment Arm 2; Mastergraft Granules (medical device made of medical grade combination of hydroxyapatite and beta-tricalcium phosphate).
Who Masked: Participant
Masking Description: This is a single-blinded study. The study participants will be blinded to the study randomisation assignment and study treatment they receive. In addition, every effort will be made by the Sponsor and Investigator to maintain the study blind. Treatment assignment will occur in sequential chronological order according to a central master list of random assignments prepared by the study statistician (master randomization list).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NeoFuse (Experimental): Anterior Cervical Discectomy and Fusion with NeoFuse.
  NeoFuseTM is constituted of STRO-3 immunological selected allogeneic MPCs, which are derived from adult bone marrow mononucleated cells that are culture-expanded and subsequently cryopreserved.
  The allogeneic MPCs are formulated in concentrations of nucleated cells in a 5 mL volume and are cryopreserved in 7.5% dimethyl sulfoxide (DMSO)/50% Alpha Modified Eagle's Medium (MEM) and 42.5% ProFreeze®. The final formulation consists of 0.15mL (approximately 10 million MPCs) of thawed NeoFuse™ thawed NeoFuseTM combined with the amount of MasterGraftTM Matrix to fill the PEEK cage per ACDF level.
  Interventions: Biological: NeoFuse
- MasterGraft Granules (Active Comparator): Anterior Cervical Discectomy and Fusion with MasterGraft Granules
  MASTERGRAFT® GRANULES are a medical-grade, polyporous resorbable ceramic hybrid composed of 15% hydroxyapatite (HA) and 85% beta-tricalcium phosphate (β-TCP). The combination of these natural bone materials provides surgeons with an osteoconductive, porous implant that improves osteointegration by allowing cells to colonize throughout the implant and optimize the bone healing process
  Interventions: Device: MasterGraft Granules

INTERVENTIONS:
Biological: NeoFuse — Single Dose NeoFuse Surgical Implantation
  Other Names: Anterior Cervical Discectomy and Fusion with NeoFuse; Cervical Spinal Fusion; Adult Stem Cells
  Arms: NeoFuse
Device: MasterGraft Granules — Single Dose MaterGraft Granules Surgical Implantation
  Other Names: Anterior Cervical Discectomy and Fusion with Granules; Cervical Spinal Fusion; Active Control
  Arms: MasterGraft Granules

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of NeoFuse in subjects with a diagnosis of degenerative disc disease (DDD) at 2 or more adjacent cervical vertebral levels between C3-C4 to C7-T1. All subjects in this study will undergo 2 or 3 level anterior cervical discectomy and fusion with Anterior Cervical Plate Fixation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, single-blinded, controlled study evaluating safety and preliminary efficacy of immunoselected, culture-expanded, nucleated, allogeneic MPCs (NeoFuse) combined with MasterGraft Matrix in a commercially available PEEK cervical Spacer compared to an active control in subjects undergoing 2 or 3 level anterior cervical discectomy and fusion with anterior cervical plate fixation.

After the screening and surgical visits, each subject will be evaluated clinically and radiographically within 3 days and 30 days after surgery, and at 3, 6, 12, and 24 months after surgery.

Subjects will be evaluated at the same time points for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females between 18 and 70 years of age, inclusive.
2. Has the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Has the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI).
4. Has a documented symptomatic diagnosis of DDD at C3-C4 to C7-T1.
5. Has symptomatic radiculopathy and/or myelopathy correlating to radiographic findings of duration of 6 weeks or greater that had failed to respond to non-operative management
6. Is a candidate for anterior cervical discectomy and fusion in two or three adjacent cervical interbody levels between C3-C4 to C7-T1
7. Has a stable screening electrocardiogram (ECG), as determined by the investigator that would not preclude surgery.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following surgery.
2. Has a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
3. Has at the time of surgery a systemic or local infection at the site of proposed surgery.
4. Has or is undergoing revision of a prior fusion surgery at any involved level.
5. Requires ACDF at only one cervical interbody level or more than 3 adjacent cervical interbody levels.
6. Requires ACDF without the use of an anterior cervical plating system.
7. Has osteoporosis as defined by a DEXA T score of ≤ -3.0 or a history of fragility fractures or other significant bone disease contraindicating the use of spinal instrumentation.
8. Has a documented medical history or radiographic evidence of a metabolic bone disease or other condition which would negatively impact the bone healing process.
9. Has a positive screen for human immunodeficiency virus (HIV) antibodies.
10. Has had treatment with any investigational therapy or device within 6 months of study surgery and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial during the 2-year follow-up period.
11. Has been a recipient of prior stem cell/progenitor cell therapy for spinal fusion surgery.
12. Has 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens.
13. Is transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety of NeoFuse | 2 years
  To determine the safety of NeoFuse using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests (hematology, serum chemistry, inflammation, and and immunology).

SECONDARY OUTCOMES:
Fusion success with NeoFuse | 1 year
  To evaluate the fusion success with NeoFuse compared to an active control using CT scans and x-ray of the involved cervical spine levels and assess the change in outcomes (NDI, SF-36, Zung Depression Questionnaire, and WPAI.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brown, Study Director — Mesoblast, Ltd.
Locations (2):
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- See also: Sponsor Website — http://www.mesoblast.com